CLINICAL TRIAL: NCT06088069
Title: Effect of Virtual Reality on Perioperative Anxiety, Stress and Pain in Total Hip Arthroplasty: a Randomized Controlled Trial
Brief Title: Effect of Virtual Reality on Perioperative Anxiety, Stress and Pain in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR331/9/23
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Virtual Reality; Total Hip Arthroplasty; Anxiety; Stress; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group VR (Experimental): Patients will be virtually immersed into a natural universe and soft music for 15 minutes preoperatively and during surgery.
  Interventions: Other: Virtual reality
- Group C (No Intervention): Patients will not receive Virtual reality (VR) experience.

INTERVENTIONS:
Other: Virtual reality — Patients will be virtually immersed into a natural universe and soft music for 15 minutes preoperatively and during surgery.
  Arms: Group VR

SUMMARY:
The aim of this study is to evaluate Virtual reality (VR) on perioperative anxiety, pain, hemodynamics, and stress hormones in patients undergoing Total hip arthroplasty (THA).

DETAILED DESCRIPTION:
VR is a computer technology that provides the feeling of being immersed in a simulated three-dimensional (3D) world where the user may interact with the virtual environment. Clinical studies have shown that VR technology is effective in reducing pain perception and anxiety. It has also been proposed as an effective non-pharmacological alternative for reducing acute procedural pain and providing anxiety relief.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or above.
* Both sexes.
* The American Society of Anesthesiologists (ASA) physical status I-III.
* Scheduled for elective THA under spinal anesthesia.

Exclusion Criteria:

* Cerebrovascular disease.
* Psychiatric-cognitive dysfunction.
* Claustrophobia.
* Deaf and blind patients.
* Uncooperative.
* Adrenal insufficiency.
* Chronic alcohol and substance addiction.
* Chronic sedative and narcotic use.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Anxiety | 15 min before operation till immediately postoperative.
  Each patient will be instructed about the scores; State Anxiety Inventory (STAI-S).
  The Arabic validated version of STAI-S test will be provided to the patients to determine the anxiety levels.
  Scores vary between and 20-80 with high scores associated with higher anxiety levels. Patients will be asked to read each statement and then indicate how they were feeling at that moment by marking the appropriate parentheses on the right side of each statement.
  Anxiety will be measured at baseline (15 min before operation), before spinal anesthesia and immediately postoperative.

SECONDARY OUTCOMES:
Total intraoperative haloperidol consumption | Intraoperatively.
  Rescue sedation (haloperidol 2.5 mg titrated doses till the needed effect) will be given if the patient is still in anxiety.
Stress measured by Cohen Perceived Stress Scale | 15 min before operation till immediately postoperative.
  Patients will be asked about feelings and thoughts during the last month to indicate how often you felt or thought a certain way on a five-point scale from 'never' to 'very often'. Answers are then scored as follow: Never=0, Almost never=1, Sometimes=2, Fairly often=3, Very often=4. It consists of 10 questions, takes 5-10 minutes to complete and is for individual or group administration.
  Stress scores will be measured at baseline (15 min before operation), before spinal anesthesia and immediately postoperative.
Stress measured by blood serum level of cortisol | 6 hours postoperative.
  Serum cortisol level will be measured before surgery and 6 h
The degree of postoperative pain | 24 hours postoperatively.
  Numerical Rating Scale(NRS) will be assessed to evaluate postoperative pain and ask patients to rate their level of pain at 30 minutes and then at 2, 4, 6, 12, 18 and 24 hours postoperative on a scale specifically adapted for this purpose. Each patient obtained a score between 0 and 10.
Amount of opioid consumption | 24 hours after surgery.
  All patients will be given paracetamol 1 g as routine analgesia. If Numerical Rating Scale (NRS) > 3 is observed, rescue analgesia (pethidine 0.5 mg IV) will be administered.
Heart rate changes | Till the end of surgery.
  Heart rate (HR) will be measured at baseline, before spinal anesthesia , and 5, 10, 15, 30, 60, 90 and 120 minutes intraoperatively and at end of surgery.
Mean arterial blood pressure changes | Till the end of surgery.
  Mean arterial blood pressure will be measured at baseline, before spinal anesthesia , and 5, 10, 15, 30, 60, 90 and 120 minutes intraoperatively and at end of surgery.
Patient satisfaction | 24 hours after surgery.
  Patient satisfaction will be assessed on a 5-point likert scale Patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied ; 5, extremely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.

REFERENCES:
- [Derived] Moharam SA, ElSharkawy MS, ELkashef AM, Romeih MA, El Rasool AOAR, Shaheen MM. Effect of virtual reality on perioperative anxiety, stress and pain in total hip arthroplasty: a randomized controlled trial. BMC Anesthesiol. 2025 Sep 9;25(1):446. doi: 10.1186/s12871-025-03316-3. PMID 40922021